CLINICAL TRIAL: NCT03866031
Title: Comparative Clinical and Radiographic Study of Mandibular Overdentures Immediately Loaded on Implants or Mini-implants Randomized Control Trial
Brief Title: Comparative Study of Mandibular Dentures Immediately Loaded on Implants or Mini-implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-RemPro-01-2019
Record Dates: First submitted 2019-03-02; First posted 2019-03-07 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Problem With Dentures
Keywords: Implant, overdenture, Immediate loading

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- M:2.75 (Experimental): 12 Patients will be provided with 4 mini implant-supported mandibular overdentures d: 2.75 mm
  Interventions: Other: implant-supported mandibular overdenture
- M3.25 (Experimental): 12 Patients will be provided with 4 mini implant-supported mandibular overdentures d: 3.25 mm
  Interventions: Other: implant-supported mandibular overdenture
- S3.75 (Experimental): 12 Patients will be provided with 2 standard sized implant-supported mandibular overdentures d: 3.75 mm
  Interventions: Other: implant-supported mandibular overdenture

INTERVENTIONS:
Other: implant-supported mandibular overdenture — The implant-supported overdentures will be placed in immediate functional loading on the same day of implants placement. A direct restorative protocol will be applied to modify the existing prosthesis to implant-supported overdentures.

SUMMARY:
3 groups of immediately Loaded implant-supported overdenture patients will be evaluated (overdentures supported by two standard-sized implant, overdentures supported by 4 mini implant d: 3.2 mm ,overdentures supported by 4 mini implant d: 2.75 mm) regarding stability, masticatory efficiency, patient's satisfaction, oral health related quality of life, Peri-implant crestal alveolar bone loss.

DETAILED DESCRIPTION:
The implant-supported overdentures will be placed in immediate functional loading on the same day of implants placement. A direct restorative protocol will be applied to modify the existing prosthesis to implant-supported overdentures.

The evaluations of the primary outcomes will be conducted before implantation and after (1 - 3 - 6 - 12 - 18), except Peri-implant crestal alveolar bone loss will be conducted only after (0 - 3 - 6 - 12 - 18).

ELIGIBILITY:
Inclusion Criteria:

1. the patient should be completely edentulous for at least 6 months.
2. first class jaw relation.
3. adequate bone for an implant length of at least 10 mm and diameter of at least 2.75 mm.
4. the patients should be able to speak and write in arabic.

Exclusion Criteria:

1) patients who received radiotherapy to the head or neck region for tumors. (2) a history of chemotherapy. (3) patients on long-term steroids, or bisphosphonates. (4) heavy smokers. (5) patients with physical and mental dis -abilities that interfere with the maintenance of implants.

(6) uncontrolled systematic disease that could compromise implant surgery. (7) extreme bruxism. (8) infectious disease. (9) temporomandibular joint dysfunction.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
change in denture stability | T1: before implantation; T2: 1 month after loaded; T3: 3 month after loaded; T4: 6 month after loaded; T5:12 month after loaded
  The evaluation will be by Digital force gauge, a Hook of orthodontic wire (18 gauge diameter) will attach to the labial flange of overdenture, the other end of wire will connect to the force gauge which will be pull vertically upward until denture retention lost, and then reading will record 3 times and means value will calculate.
change in masticatory efficiency | T1: before implantation; T2: 1 month after loaded; T3: 3 month after loaded; T4: 6 month after loaded; T5:12 month after loaded
  The evaluation will be by test food filtering device,Where the subjects will chew a measured portion of test food (peanuts) for 20 strokes. The test food will strain through mesh sieve (2 mm opening). The volume of food remaining on the sieve and that passing through the sieve determined the masticatory performance.
change in patient's satisfaction | T1: before implantation; T2: 1 month after loaded; T3: 3 month after loaded; T4: 6 month after loaded; T5:12 month after loaded
  The evaluation will be by 100 mm Visual Analog Scale (VAS), for which higher scores indicate greater satisfaction, They will be asked to rate their level of comfort, ability to chew, stability, ability to speak, ease of cleaning their prostheses and their general satisfaction.
change in oral health related quality of life | T1: before implantation; T2: 1 month after loaded; T3: 3 month after loaded; T4: 6 month after loaded; T5:12 month after loaded
  The evaluation will be by oral health impact profile of edentulous (Ohip-Edent) instrument, Patients will answer questions of ohip-edent which included 7 domains: functional limitation, physical pain, psychological discomfort, physical disability, Psychological disability, Social disability, Handicap. Responses will made on a five-grade Likert-type scale:
  0=never ; 1=hardly ever ; 2=occasionally ; 3= fairly often ; 4= very often. disability, social disability and handicap
change in Peri-implant crestal alveolar bone loss | T1: on same day of loaded; T2: 3 month after loaded; T3: 6 month after loaded; T4:12 month after loaded
  The evaluation will be by panoramic radiogram, Peri-implant vertical and horizontal alveolar bone loss will measure (in mm) at the mesial and distal surface of each implant.
  implant

CONTACTS AND LOCATIONS:
Overall Officials: Heba M Moftah, DDS MSc, Principal Investigator — PhD student at Removable Prosthodontics Department, faculty of dental medicine, Damascus Univ; Mohannad H Al-saadi, DDS MSc PhD, Study Director — Professor of Removable Prosthodontics, faculty of dental medicine, Damascus Univ; Khaldoun A Darwich, DDS Msc PhD, Study Director — Professor of Oral and Maxillofacial surgery, faculty of dental medicine, Damascus Univ
Locations (1):
- Removable prosthodontics department and implantation department / Faculty of dental medicine / Damascus univ, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zygogiannis K, Aartman IH, Parsa A, Tahmaseb A, Wismeijer D. Implant Mandibular Overdentures Retained by Immediately Loaded Implants: A 1-Year Randomized Trial Comparing the Clinical and Radiographic Outcomes Between Mini Dental Implants and Standard-Sized Implants. Int J Oral Maxillofac Implants. 2017 Nov/Dec;32(6):1377-1388. doi: 10.11607/jomi.5981. PMID 29140382
- [Background] Kanazawa M, Tanoue M, Miyayasu A, Takeshita S, Sato D, Asami M, Lam TV, Thu KM, Oda K, Komagamine Y, Minakuchi S, Feine J. The patient general satisfaction of mandibular single-implant overdentures and conventional complete dentures: Study protocol for a randomized crossover trial. Medicine (Baltimore). 2018 May;97(20):e10721. doi: 10.1097/MD.0000000000010721. PMID 29768340
- [Background] ALHarthi SS, BinShabaib MS, Ahmed HB, Mehmood A, Khan J, Javed F. Comparison of peri-implant clinical and radiographic inflammatory parameters among cigarette and waterpipe (narghile) smokers and never-smokers. J Periodontol. 2018 Feb;89(2):213-218. doi: 10.1902/jop.2017.170358. PMID 28777038
- [Background] Kappel S, Giannakopoulos NN, Eberhard L, Rammelsberg P, Eiffler C. Immediate Loading of Dental Implants in Edentulous Mandibles by Use of Locator(R) Attachments or Dolder(R) Bars: Two-Year Results from a Prospective Randomized Clinical Study. Clin Implant Dent Relat Res. 2016 Aug;18(4):752-61. doi: 10.1111/cid.12349. Epub 2015 May 7. PMID 25950679
- [Background] Kroll P, Hou L, Radaideh H, Sharifi N, Han PP, Mulligan R, Enciso R. Oral Health-Related Outcomes in Edentulous Patients Treated With Mandibular Implant-Retained Dentures Versus Complete Dentures: Systematic Review With Meta-Analyses. J Oral Implantol. 2018 Aug;44(4):313-324. doi: 10.1563/aaid-joi-D-17-00210. Epub 2018 Feb 19. PMID 29457932